CLINICAL TRIAL: NCT04555200
Title: Continuous Enteral Rehydration by Nasogastric Tube With ORS in Children With Acute Gastroenteritis: Evaluation of Professional Practices Before and After Protocol Change
Brief Title: Continuous Enteral Rehydration by Nasogastric Tube With ORS in Children With Acute Gastroenteritis
Acronym: GEA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0130
Record Dates: First submitted 2020-07-06; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2019-09

CONDITIONS: Acute Gastroenteritis; Dehydration
Keywords: nasogastric tube; Emergency medicine; Pediatric medicine
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When oral rehydration is impossible, enteral rehydration via the nasogastric route has been the recommended method of rehydration since 2008 by ESPGHAN ( European Society for Paediatric Gastroenterology Hepatology and Nutrition ), for children with acute gastroenteritis. However, these recommendations are rarely followed in France. These recommendations were not applied in the Children's Emergency Department of BREST University Hospital. The investigators changed the protocol and shared it with the caregivers of the emergency unit. The investigators studied the impact of this change of protocol

DETAILED DESCRIPTION:
The main purpose was to assess the proportion of children rehydrated by nasogastric tube(NG) after protocol change. Secondary outcomes were to assess hospital length of stay and sides effects.

It is a retro and prospective study. The first phase took place from June to September 2018 and the second from June to September 2019. Any child presenting to pediatric emergencies for acute gastroenteritis requiring nonoral rehydration was included.

ELIGIBILITY:
Inclusion Criteria:

Any child presenting to pediatric emergencies for acute gastroenteritis requiring nonoral rehydration was included

Exclusion Criteria:

* acute gastroenteritis on return from tropical countries
* child with endocrine system diseases requiring parenteral rehydration
* history of chronic pathology requiring enteral feeding

Ages: 1 Day to 15 Years | Sex: All
Age Groups: Child
Study Population: Any child from 0 to 15 years presenting to pediatric emergencies for acute gastroenteritis requiring nonoral rehydration was included
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Number of nasogastric tube after changing gastroenteritis rehydration protocol | 4 months
  assessed by the number of NG tube and IV in each group

SECONDARY OUTCOMES:
Hospital lenght of stay between each group | 4 months
  evaluate by administrative data of each case (arrival time and departure time)
Number of Participants With Treatment-Related Adverse Events for each method | 4 months
  Serious sides effect were death and epilptic seizure. Mild sides effects were multiple (IV or NG ripped out, vomiting, failure...).

CONTACTS AND LOCATIONS:
Overall Officials: Nadege Delaperriere, Doctor, Principal Investigator — CHRU Brest
Locations (1):
- CHRU de Brest (urgences pédiatriques), Brest, France